CLINICAL TRIAL: NCT02353390
Title: Feasibility and Impact of Implementing an Oral Water Hydration Strategy to Prevent Post-Vaccination Presyncope and Syncope in Adolescents and Young Adults
Brief Title: Oral Water Hydration to Prevent Post-Vaccination Presyncope
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Duke University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Boston University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: Pro00060114; 200-2012-53663 0005 (Other Grant/Funding Number: Centers for Disease Control and Prevention)
Record Dates: First submitted 2015-01-28; First posted 2015-02-02 (Estimated); Last update posted 2016-07-07 (Estimated); Status verified 2016-06

CONDITIONS: Presyncope; Syncope
Keywords: presyncope; syncope; adolescent; young adult; immunization; vaccination; water consumption
MeSH Terms: conditions — Syncope

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Oral Water Hydration (Active Comparator): Subjects will be given up to 15 minutes to drink up to 500 mL of water prior to the first IM vaccination.
  Interventions: Other: Oral Water Hydration
- Usual Care (No Intervention): Subjects will receive usual care prior to the first IM vaccination. No water or food will be offered.

INTERVENTIONS:
Other: Oral Water Hydration — Subjects in the hydration group will be allowed up to 15 minutes to drink up to 500 milliliters (mL) of water prior to the vaccines. Subjects will be encouraged to drink the entire 500 mL; however, they are free to drink as much as they want and can finish before the end of the 15-minute period. Subjects will be instructed not to share the water and to not otherwise empty the bottle. As with the control group, subjects will be instructed not to eat or drink anything else for the duration of the study, unless clinically indicated (e.g., as part of management of presyncope or syncope).
  Arms: Oral Water Hydration

SUMMARY:
This is a randomized controlled open-label trial. During the study, adolescents and young adults scheduled to receive at least one intra-muscular (IM) vaccine will receive either oral water hydration in addition to standard care or standard of care alone to evaluate the effect of water hydration on the primary outcome of presyncope. This study will also evaluate the acceptability of pre-vaccination hydration among adolescents and young adults.

DETAILED DESCRIPTION:
Post-vaccination syncope is a rare but potentially serious adverse event in adolescents and young adults. Because few data are available regarding post-vaccination syncope, evidence regarding presyncope and syncope after blood donation provides useful insight. Based on studies of blood donors, acute water loading fifteen minutes prior to vaccination with 500 mL of water might reduce the risk of syncope. However, the degree to which hydration attenuates the risk of post-vaccination syncope or presyncope is unknown. Furthermore, little is known about the acceptability of pre-vaccination hydration to adolescents and young adults.

The objective of this study is to conduct a study to evaluate the acceptability and impact of oral hydration to prevent presyncope following vaccination in adolescents and young adults 11 through 21 years of age. The primary objectives are to determine if pre-vaccination hydration decreases the rate of presyncope in adolescents and young adults receiving at least one intra-muscular (IM) vaccine and to determine if pre-vaccination hydration is acceptable to adolescents and young adults.

This is a randomized controlled open-label study in adolescents and young adults receiving at least one IM vaccine. Vaccine administration will be part of routine care and will not be a study procedure. Adolescents and young adults 11- through 21 years of age will be eligible for participation. Minimal subject exclusion criteria will be used to best reflect how pre-vaccination hydration could be used outside of the controlled trial setting. For all primary and secondary objectives, data will be collected before and after vaccination, with data collection to be completed on the day of enrollment.

ELIGIBILITY:
Inclusion Criteria:

* The subject must be 11 years through 21 years of age
* The subject must be receiving at least one IM vaccine
* If the subject is younger than 18 years and not able to give independent consent under the applicable laws of the local jurisdiction, the parent/guardian must be willing and capable of providing written informed consent for the child and the child must be willing and capable of providing assent OR if the subject is 18 years or older or younger than 18 years and able to give independent consent under the applicable laws of the local jurisdiction, the subject must be willing and capable of providing written informed consent.
* The subject must be willing to stay for the completion of all study-related activities.
* The subject must be willing to try to drink up to 500 ml water in a pre-specified period of time (15 minutes) prior to receipt of prescribed vaccines.

Exclusion Criteria:

* No experimental vaccine or medication within the previous two weeks
* No daily injectable medication
* No permanent indwelling venous catheter
* No blood drawn within the past hour or scheduled for a blood draw during the post-vaccination observation period
* Any condition that would, in the opinion of the site investigator, place the participant at an unacceptable risk of injury or render the participant unable to meet the requirements of the protocol

Ages: 11 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 1820 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Presyncope | 20 minutes
  Sudden onset of one or more of the following symptoms or signs during the post-vaccination observation period in the clinic:
  Symptoms
  * Feeling lightheaded, like you might "pass out" or faint
  * Feeling dizzy, like the room is spinning
  * Feeling weak
  * Feeling like your face is getting red and warm (or hot), like blushing
  * Noticing any change in your vision, like spots or flickering lights, tunnel vision, or loss of vision
  * Experiencing ringing in your ears, decreased hearing, or sounds seem far away
  * Feeling like your heart is beating fast or hard or pounding
  * Feeling hot AND sweaty
  * Feeling cold AND sweaty, or "clammy"
  * Feeling like you are breathing fast or hard
  * Feeling like you might throw up (nausea)
  Signs
  * Pallor
  * Sweaty
  * Facial flush
  * Decreased interactivity (decreased level of arousal or responsiveness)
  AND
  * Not Syncope
  * Not due to another cause
  * Not clearly present at baseline
Acceptability of oral water hydration in the intervention group, assessed by qualitative reports in the post-vaccination observation period and response to a survey about whether they liked getting water. | 20 minutes

SECONDARY OUTCOMES:
Syncope | 20 minutes
  Syncope (fainting) that occurs in an otherwise healthy person after receipt of a vaccine or during venipuncture is usually attributed to vasovagal syncope, and may occur alone (simple syncope) or may be associated with tonic-clonic movements (convulsive syncope, anoxic seizure). For the purposes of this study, we have defined syncope as: Any sudden and brief loss of consciousness or postural tone after vaccination from which recovery is spontaneous and is not attributed to another cause (e.g., anaphylaxis). For purposes of this study, cases counted as syncope must occur during the post-vaccination observation period.
  Individuals that develop syncope after presyncope will be classified only as having syncope.
Alternative Case Definition of Presyncompe | 20 minutes
  In secondary analysis, the case definition of presyncope (Outcome 1) will be defined as any response of self-report of the symptoms of presyncope at a level of "somewhat," "a lot," or "extremely" compared to "none" or "a little."

CONTACTS AND LOCATIONS:
Overall Officials: Alex R Kemper, MD, MPH, MS, Principal Investigator — Duke University; Elizabeth D Barnett, MD, Principal Investigator — Boston University; Theresa Harrington, MD, Principal Investigator — Centers for Disease Control and Prevention
Locations (2):
- United States (2):
  - Boston Medical Center, Boston, Massachusetts
  - Duke University Medical Center, Durham, North Carolina

REFERENCES:
- [Background] Braun MM, Patriarca PA, Ellenberg SS. Syncope after immunization. Arch Pediatr Adolesc Med. 1997 Mar;151(3):255-9. doi: 10.1001/archpedi.1997.02170400041007. PMID 9080932
- [Background] National Center for Immunization and Respiratory Diseases. General recommendations on immunization --- recommendations of the Advisory Committee on Immunization Practices (ACIP). MMWR Recomm Rep. 2011 Jan 28;60(2):1-64. PMID 21293327
- [Background] Centers for Disease Control and Prevention (CDC). Syncope after vaccination--United States, January 2005-July 2007. MMWR Morb Mortal Wkly Rep. 2008 May 2;57(17):457-60. PMID 18451756
- [Background] Hanson SA, France CR. Predonation water ingestion attenuates negative reactions to blood donation. Transfusion. 2004 Jun;44(6):924-8. doi: 10.1111/j.1537-2995.2004.03426.x. PMID 15157261
- [Background] Newman B, Tommolino E, Andreozzi C, Joychan S, Pocedic J, Heringhausen J. The effect of a 473-mL (16-oz) water drink on vasovagal donor reaction rates in high-school students. Transfusion. 2007 Aug;47(8):1524-33. doi: 10.1111/j.1537-2995.2007.01293.x. PMID 17655598
- [Background] Soteriades ES, Evans JC, Larson MG, Chen MH, Chen L, Benjamin EJ, Levy D. Incidence and prognosis of syncope. N Engl J Med. 2002 Sep 19;347(12):878-85. doi: 10.1056/NEJMoa012407. PMID 12239256